CLINICAL TRIAL: NCT04347512
Title: EVALUATION OF THE EFFICACY OF THE HYDROXYCHLOROQUINE-AZITHROMYCIN COMBINATION IN THE IN THE PREVENTION OF COVID-19 RELATED SDRA
Acronym: TEACHCOVID
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: In view of the notices concerning hydroxychloroquine issued by the regulatory authorities, we withdraw the protocol
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7783
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Sars-CoV-2, Community-Acquired Pneumonia,COVID-19
MeSH Terms: conditions — Community-Acquired Pneumonia; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine (Experimental): Hydroxychloroquine is given for 5 days, with a loading dose of 400 mg qd at D1, and 200 mg qd for the next 4 days (D2-D5).
  Standard of care is also prescribed (oxygen therapy, analgesics, antipyretics, anticoagulant drug, etc)
  Interventions: Drug: Hydroxychloroquine
- Control (Active Comparator): The patient is given antibiotics only. Standard of care is also prescribed (oxygen therapy, analgesics, antipyretics, anticoagulant drug, etc).
  Interventions: Drug: Control arm
- Hydroxychloroquine and Azithromycin (Experimental): Hydroxychloroquine is given for 5 days, with a loading dose of 400 mg qd at D1, and 200 mg qd for the next 4 days (D2-D5).
  Azithromycin is given for 5 days, with a loading dose of 500 mg at D1, and 250 mg for the next 4 days.
  Standard of care is also prescribed (oxygen therapy, analgesics, antipyretics, anticoagulant drug, etc) In case of moderate renal failure (glomerular filtration rate between 30 and 60 mL/min/m²), hydroxychloroquine dosage are lowered by half.
  Interventions: Drug: Hydroxychloroquine and azithromycin treatment arm.

INTERVENTIONS:
Drug: Hydroxychloroquine and azithromycin treatment arm. — Patient allocated in this arm receive hydroxychloroquine and azithromycin for 5 days.
  For hydroxychloroquine, there is a loading dose of 800 mg per day at D1, followed by 400 mg per day D2-D5.
  For azithromycin, there is a loading dose of 500 mg per day at D1, followed by 250 mg per day D2-D5.
  Every patient receive as well antibiotic (ceftriaxone 1-2 g per day IV), and standard of care (oxygen therapy, analgesics, antipyretics, heparin, etc).
  Arms: Hydroxychloroquine and Azithromycin
Drug: Hydroxychloroquine — Patient allocated in this arm receive hydroxychloroquine for 5 days. For hydroxychloroquine, there is a loading dose of 800 mg per day at D1, followed by 400 mg per day D2-D5.
  Every patient receives as well antibiotic (ceftriaxone 1-2 g per day IV), and standard of care (oxygen therapy, analgesics, antipyretics, heparin, etc).
  Arms: Hydroxychloroquine
Drug: Control arm — In this arm, no experimental treatment is prescribed. Patients receive IV antibiotics and standard of care (oxygen therapy, analgesics, antipyretics, heparin, etc).
  Arms: Control

SUMMARY:
Since end of December, a new coronavirus, close to the 2002 SARS coronavirus, cause serious pneumonias throughout world. There is currently no strong evidence of an efficient specific treatment. Hydroxychloroquine is an old chloroquine-derived drug, prescribed for auto-immune disorders. It has shown efficacy against Sars-CoV-2 in vitro. Some studies showed that Hydroxychloroquine might improve the clinical status of Sars-CoV-2 infected patients. Azithromycin is a macrolide antibiotic, with immunomodulatory properties. Adding Azithromycin to a hydroxychloroquine-based treatment showed an apparent accelerated viral clearance in infected patients. This study wants to evaluate the clinical impact of adding Azithromycin to Hydroxychloroquine in the treatment of Sars-CoV-2 pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Positive Sars-CoV-2 RT-PCR on nasopharyngeal swab
* CT scan suggestive of Sars-CoV-2 pneumonia

Exclusion Criteria:

* Negative Sars-CoV-2 RT-PCR on nasopharyngeal swab
* Known hypersensitivity to Hydroxychloroquine, Azithromycin or a macrolide family member
* Long term prescribed treatment contraindicated with azithromycin (colchicine, ergotamine, dihydroergotamine) and/or hydroxychloroquine (citalopram, escitalopram, hydroxyzine, domperidone, piperaquin)
* Retinopathy or maculopathy
* Porphyria
* Severe renal failure (GFR less than 30 mL/min/m²)
* Dyskaliemia, (ie less than 3,5 mmol/L or more than 5,5 mmol/L)
* Hypomagnesiemia, ie less than 0,7 mmol/L
* Severe cholestasis, cirrhosis or severe hepatic failure
* Known cardiac medical history of congestive heart failure or myocardial infarction
* Bradycardia less than 50 beats per minute
* Prolonged corrected QT interval, (ie cQT more than 440 ms in men and 450 ms in women) or medical history of ventricular cardiac rhythm disorders
* Blood disorders with history of hematopoietic stem cells allograft
* Known history of G6PD deficiency
* Pregnancy
* Breastfeeding
* Subject protected by law under guardianship of curatorship
* Inability to take oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Rate of patients reaching a significant hypoxemia, in each arms. | From day 0 to day 7
  A significant hypoxemia is an arterial partial pressure of oxygen of less than 60 mmHg despite an oxygen flow of more than 6 L/min, patient at rest.

IPD SHARING:
Plan to Share IPD: No